CLINICAL TRIAL: NCT01199341
Title: A Phase I, Open Label, Randomised, Parallel Group Study of Repeated Oral Doses of AZD1981 (100 mg Twice Daily and 400 mg Twice Daily) for Two Weeks and Single Doses of Warfarin (25 mg) to Evaluate the Pharmacokinetic Interaction of AZD1981 and Warfarin and the Effect of AZD1981 on Warfarin Pharmacodynamics in Healthy Male Volunteers
Brief Title: A Drug-Drug Interaction Study to Study the Effect of AZD1981 on Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D9830C00017; 2010-021956-24 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Pharmakokinetic
Keywords: Phase 1; Drug-Drug interaction; warfarin; AZD1981
MeSH Terms: interventions — AZD1981; Warfarin; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): AZD1981, low dose, + Warfarin
  Interventions: Drug: AZD1981; Drug: Warfarin
- Treatment B (Experimental): AZD1981, high dose, + Warfarin
  Interventions: Drug: Warfarin; Drug: AZD1981

INTERVENTIONS:
Drug: AZD1981 — 100 mg per oral, twice daily for 14 days
  Arms: Treatment A
Drug: Warfarin — 10 x 2.5 mg per oral, once daily at day 1 and day 15
  Other Names: Waran
Drug: AZD1981 — 4 x 100 mg per oral, twice daily for 14 days
  Arms: Treatment B

SUMMARY:
The primary purpose of this study is to determine whether the treatment with AZD1981 affect the exposure of Warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index between 19 and 30 kg/m2 and weight at least 65 kg and no more than 100 kg
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to screening
* Volunteers must be willing to use barrier methods of contraception during study and 3 months after the end of their participation in the study

Exclusion Criteria:

* Volunteer that is inferred to have an increased sensitivity to warfarin based on genotype of CYP2C9 and VKORC1.
* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings in physical examination

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics for (R)- and (S)-Warfarin, respectively measured by Cmax and Area Under the Curve (AUC) | PK sampling will be performed regularly from Day 1 to Day 22

SECONDARY OUTCOMES:
Explore possible changes in the anticoagulative activity of Warfarin measured by INR . | Will be performed at screening and at all visits during the study period.
Pharmacokinetics for AZD1981 measured by AUCτ, Css,max, tmax,ss and CLss/F | PK sampling will be performed regularly from Day 15 to Day 22.
Safety and tolerability of AZD1981 | Safety will be monitored continuously and safety assessments will be made on several occasions throughout the whole study.

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultqvist, MD, Study Director — AstraZeneca; Aslak Rautio, Principal Investigator — Quintiles AB; Wofgang Kühn, MD, Principal Investigator — Quintiles AB
Locations (1):
- Research Site, Uppsala, Sweden